CLINICAL TRIAL: NCT03082859
Title: A Comparison of the Acute Impact of High-intensity Interval Training, Reduced-exertion High-intensity Interval Training and Moderate-intensity Continuous Aerobic Exercise on Free-living Glycaemic Control in Type 2 Diabetes
Brief Title: Acute Exercise and Free-living Glycaemic Control in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Diabetes Research and Wellness Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16/NI/0115
Record Dates: First submitted 2016-08-12; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: Exercise; Interval Training; Glycaemic Control; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Reduced-exertion high-intensity interval training (Experimental): Cycling Exercise. 2 x 20-sec sprints.
  Interventions: Behavioral: Exercise
- High Intensity Interval Training (HIT) (Experimental): Cycling Exercise. 10 x 1 min at approx 85% peak power output (Wmax)
  Interventions: Behavioral: Exercise
- Moderate Intensity Continuous Exercise (Experimental): Cycling exercise. 30 min at 50% peak power output (Wmax)
  Interventions: Behavioral: Exercise
- Sedentary (no exercise) (No Intervention): No exercise. Rest.

INTERVENTIONS:
Behavioral: Exercise — This a randomised cross-over study involving three different modes of exercise which will be compared to a no-exercise control.
  Arms: High Intensity Interval Training (HIT); Moderate Intensity Continuous Exercise; Reduced-exertion high-intensity interval training

SUMMARY:
Exercise is considered one of the three cornerstones of type 2 diabetes (T2D) care programmes (together with diet and medication), yet the majority of individuals with T2D do not achieve the minimum recommended levels of physical activity. Two of the key barriers to exercise appear to be a 'lack of time' and the high levels of perceived exertion and fatigue. At Ulster University, it has recently been demonstrated that a modified high-intensity interval training (HIT) intervention, consisting of 10-min of low-intensity cycling interspersed with two 20-s 'all-out' sprints (reduced-exertion HIT; REHIT), was effective at improving insulin sensitivity in sedentary men over six weeks. Importantly, these benefits were observed despite the very low time commitment (just 10-min per session) and relatively low ratings of perceived exertion ('somewhat hard'). As REHIT is associated with substantial muscle glycogen breakdown, we hypothesise that this exercise mode may also acutely improve glycaemic control in patients with T2D. This study will:

1. Examine the acute impact of REHIT, compared with a no-exercise control, on 24-hour glycaemic control under dietary-controlled but otherwise 'free-living' conditions using continuous glucose monitoring.
2. Compare the effects of REHIT with currently recommended levels of aerobic exercise and a previously recommended HIT model, both of which have been shown to improve 24-hour glycaemic control in T2D.
3. Collect information on individual's perceptions of each exercise mode through measures of affect, motivation, perceived exertion, fatigue, enjoyment and attentional focus.

DETAILED DESCRIPTION:
This study aims to determine the effects of a novel high-intensity interval exercise session (REHIT) on blood glucose levels over a typical 24 hour period. The effects of REHIT will be compared with another form of high intensity interval exercise that has previously been shown to be beneficial in T2D and with currently recommended moderate intensity aerobic exercise.

Participants:

21 men (aged 18-60) with type 2 diabetes will be recruited. Volunteers will be eligible to take part if they have been diagnosed with type 2 diabetes by a clinician at least 3 months prior to the study, and do not have any of the exclusion criteria for the study. Potential volunteers will be checked for reasons why the strenuous exercise may be unsuitable for them. Participants will be informed of the experimental protocol, and potential risks, both verbally and in writing before providing their written informed consent. The study will be conducted in accordance with the Declaration of Helsinki.

Pre-Screening and Baseline testing:

Before examining the effects of exercise participants will be asked to come to the lab on 5 separate occasions, which will be arranged to accommodate individual schedules:

1. First an electrocardiography (ECG) test will be performed to assess the function of the participants heart at rest and during exercise. This would be conducted, monitored and reviewed by a trained cardiac physiologist and involves the attachment of several small sticky pads (with wire attachments) across the chest which will measure the electrical activity in the heart. This will be done firstly at rest and then participants will be asked to cycle on a stationary bike, with the exercise intensity slowly getting harder and harder until they can't go any further.
2. Participants will then come to come to the lab after an overnight fast for collection of a fasting venous blood sample. This sample will be collected be a trained phlebotomist and will be used to measure fasting blood glucose and HbA1c for participant characterisation purposes.
3. A cycling fitness test will then be performed. For this test participants will be asked to cycle on a stationary bike, with the exercise intensity slowly getting harder and harder until you can't go any further. This test will normally take no longer than ~10 minutes but they will be in the lab for approximately 60 minutes. We will measure the maximal amount of oxygen the participant can use (a good indicator of fitness) by asking them to breathe through a mouth-piece connected to an oxygen analyser.
4. During the fourth and fifth visits participants will be given the opportunity to try out the exercise sessions that we will use in the main study, in order to get a 'feel' for what they will be asked to do. These sessions will take less than half an hour each.

Main Experimental Trials:

Participants will complete four main experimental trials which will each take place over a period of 3 days. During each trial we will measure the effects of a different type of exercise on blood glucose levels over a ~42-hour period (6pm on DAY1 until 12pm on DAY3). Participants will be provided with all meals and drinks during this period and will ask them to eat them at the same time of day during each trial. Each of these trials will be separated by at least 5 days and before each trial and participants will be asked to avoid any strenuous or tiring physical activities for 3 days. Over these 3 days, and for the duration of each trial, we will also ask participants to wear a small physical activity monitor. This device is a sophisticated form of heart rate monitor which also measures movement (Actiheart™) and will give us some detailed information on participants physical activity levels during each trial. This device connects to your skin either just above or below the left your chest via two adhesive pads, which can easily be detached/reattached while away from the laboratory whenever necessary (e.g., while bathing or showering). The Actiheart™ physical activity monitors are very small and comfortable to wear, and will not interfere with normal daily activities.

Participants will then attend the exercise laboratory (Magee Campus, Derry/Londonderry) between 4pm and 6pm on DAY1 so that the small glucose monitor can be fitted. Participants can then return home but will be given a standardised evening meal to be eaten at 8pm. On DAY2, we will ask participants to return the lab at 7am (after an overnight fast) where they will be provided with breakfast and then they will complete an exercise session ~1 hour later (i.e. 8:30 am). During the no-exercise trial participants will remain seated at rest during the exercise period. Participants will remain in the lab for ~45 minutes allowing the research team to monitor recovery and also complete some questionnaires relating to fatigue/tiredness as well as the enjoyment of each exercise. A short interview will also be conducted to find out about what participants thought about during each exercise session. From 09:30 am onwards participants will be able to return to their normal daily routine outside the laboratory, but will be provided with meals, snacks and drinks to be consumed at standard times until 12pm on DAY3.

Continuous Measurement of Blood Glucose:

Blood glucose levels will be measured continuously during each trial by fitting a small glucose monitor to the outside of the abdomen. This will provide information about how the body (blood glucose) responds to each meal consumed during this time period. This glucose monitor will be fitted using an automated insertion device with a short needle to insert a glucose sensor attached to a small recorder (the small needle is then immediately removed). The device itself is waterproof but additional dressings will be provided to apply while bathing or showering. Over the 42-hour measurement period the device needs to be calibrated eight times using finger-prick blood samples and a handheld blood glucose meter. This is in order to get accurate readings from the device. Two of these samples will be taken at the laboratory, but we will ask participants to take the handheld blood glucose meter home and perform the other six finger-prick measurements themselves. The procedure for this is very straightforward and is routinely performed by type 2 diabetics. All participants will be shown the procedure for obtain and finger prick blood sample and measuring blood glucose in this way.

Exercise Bouts:

The effects of three different types of exercise on blood glucose levels will be compared: 1) High-intensity interval training (HIT); reduced-exertion high-intensity interval training (REHIT); and 3) moderate intensity continuous exercise (MICE). The HIT exercise consists of ten, one-minute high-intensity intervals with one-minute of low-intensity recovery in between. The REHIT session consists of 10 minutes of very easy cycling, but with two 20-second 'all-out' sprint efforts after 3 and 6 minutes. The moderate intensity aerobic exercise will consist of 30-minutes of cycling at a moderate intensity. A fourth 'control' condition in which participants will do no exercise will also be performed. All of the exercise bouts will be performed in the exercise laboratory at Ulster University. During each exercise session information will be collected on perceptions of exertion, fatigue and enjoyment using standard questionnaires and rating scales. Heart rate will be measured continuously during each exercise session.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 year-old men who have been diagnosed with Type 2 diabetes by a clinician at least 3 months prior to the start of the study according to standard criteria.
* Able and willing to safely comply with all study procedures.
* Able to provide written informed consent whilst acknowledging their freedom to withdraw at any point during the study.
* Inactive or moderately physically active according to the International Physical Activity Questionnaire.

Exclusion Criteria:

* Aged < 18 years or > 60 years
* Female
* Insulin therapy
* Use of more than two antidiabetic drugs
* Use of βblockers
* Use of inhaled steroids (e.g. for asthma)
* Any cardiovascular condition with the exception of well-controlled uncomplicated hypertension (systolic >160 mmHg and/or >90mmHg after at least 5 min of seated rest), which is treated with no more than two drugs (either an ACE, ARB, calcium channel blocker, or diuretic)
* Cerebrovascular disease including previous stroke or aneurysm
* History of exercise-induced asthma
* History of Type 1 diabetes mellitus or a history of ketoacidosis
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug or chemical-induced, and post organ transplant)
* Any prior history of malignancy with the exception of: basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has been recurrence free for 5 years, other malignancies (regardless of site) that have been recurrence free for 10 years.
* History of respiratory disease including pulmonary hypertension or chronic obstructive pulmonary disease
* History of musculoskeletal or neurological disorders
* Active inflammatory bowel disease
* History of renal disease
* Other metabolic diseases, including hyper/ hypo parathyroidism, hyper/hypo thyroidism, and Cushing's disease.
* BMI>35 kg/m2
* Uncontrolled hypertension (systolic blood pressure >160 mm Hg and/or diastolic blood pressure >90 mm Hg after at least a 5 minute seated rest at the screening visit).
* A clinically significant resting and/or exercise ECG abnormality at the pre-screening visit which in the opinion of the cardiovascular physiologist exposes the participant to risk by take part in the main trial. In line with The Society for Cardiological Science & Technology recommendations for exercise testing, this includes:

  * Central nervous system symptoms (e.g. ataxia, dizziness, or near syncope)
  * Signs of poor perfusion (cyanosis or pallor)
  * Any detection of arrhythmias
  * Rapid ST elevation with or without pain
  * Systolic blood pressures >230mmHg
  * >2mm ST elevation with symptoms
  * >3mm ST depression without symptoms
* 'Yes' to any questions on a standard physical activity readiness questionnaire (PARQ)
* Classification as highly physically active on the International Physical Activity Questionnaire (IPAQ)
* Current participation in another research study
* Inability to fully understand the verbal and written descriptions of the study in English, and the instructions provided during the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour blood glucose concentrations (mmol/L) | 24-hours
  24-hour glucose levels will be measured with continuous glucose monitors under standard dietary conditions. Mean blood glucose (mmol/L) will be calculated.

SECONDARY OUTCOMES:
Time spent in hyperglycaemia (% of 24-h day) | 24-hours
  24-hour glucose levels will be measured with continuous glucose monitors under standard dietary conditions. The % of the day spent above 10 mmol/L will be calculated.
Incremental Area Under the Curve (AUC) | 24 Hours
  24-hour glucose levels will be measured with continuous glucose monitors under standard dietary conditions. The incremental area under the curve for the glucose response will be calculated.
Glycaemic Variability (Glucose levels) | 24-hours
  24-hour glucose levels will be measured with continuous glucose monitors under standard dietary conditions. The variability of glucose levels over the course of the day will be assessed.

OTHER OUTCOMES:
Ratings of perceived exertion (RPE) (Borg Scale) | 1 Hour
  Ratings of perceived exertion (RPE) (Borg Scale) will be collected during each exercise (at minutes corresponding to each 10% stage of the different exercise bouts; 10%, 20% etc; i.e., for up to 30 minutes of exercise). A session RPE score will then be collected using the 15-point Borg Scale 30-minutes post exercise.
Exercise Enjoyment assessed using the exercise enjoyment scale | 30 minutes
  Exercise enjoyment will be assessed using the exercise enjoyment scale immediately after each exercise bout.
Perceptions of physical tiredness and fatigue assessed using 100-mm visual analogue scale | 1 Hour
  Perceptions of physical fatigue and tiredness will be assessed using 100-mm visual analogue scales with standardised descriptors and will be assessed before, and then 0, 10, 20 and 30 minutes post-exercise. With exercise and recovery this will take approx 1-hour for each exercise condition.
Affect measured using the one-item feeling scale | 1 Hour
  During exercise psychological affect will be measured using the one-item feeling scale. This will be measured at minutes corresponding to each 10% stage of the exercise bout completed (after 10%, 20% etc of the exercise bout; i.e. for up to 30 minutes of exercise). Measures will also be taken 10, 20 and 30 minutes post-exercise. In total this measure - including exercise and recovery - will take approx. 1-hour.
Affect measured using the positive and negative affect scale (PANAS) | 30 minutes
  Changes in positive and negative affect as a result of the exercise bouts will be measured using the positive and negative affect scale (PANAS). This will be measured pre and immediately post exercise.
Mood measured using the Brunel Scale of Mood States (BRUMS) | 30 minutes
  Changes in mood states as a result of the exercise bouts will be measured using the Brunel Scale of Mood States (BRUMS). This will be measured pre and immediately post exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Metcalfe, PhD, Principal Investigator — Lecturer in Exercise and Health
Locations (1):
- Ulster University, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No